CLINICAL TRIAL: NCT01535937
Title: The Effect of Brief Potent Glutamatergic Modulation on Cocaine Dependence
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: An analysis demonstrated that running the final participants was unnecessary.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elias Dakwar, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #6403/7339R; 1K23DA031771-01 (NIH)
Record Dates: First submitted 2011-12-29; First posted 2012-02-20 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): 0.5 mg/kg of ketamine IV over 40 minutes
  Interventions: Drug: Ketamine
- midazolam (Active Comparator): 0.025 mg/kg IV over 40 minutes
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — 0.5 mg/kg IV over 40 minutes
  Other Names: ketamine 0.5 mg/kg
  Arms: Ketamine
Drug: Midazolam — 0.025 mg/kg IV over 40 minutes
  Other Names: midazolam 0.025 mg/kg
  Arms: midazolam

SUMMARY:
This project will evaluate the effect of a single sub-anesthetic dose of ketamine on the time to first cocaine use and abstinence rates in 60 treatment-seeking cocaine-dependent individuals receiving mindfulness-based relapse prevention (MBRP) therapy, using a 5 week combined laboratory-inpatient and outpatient double-blind, randomized, controlled trial.

DETAILED DESCRIPTION:
he study will begin with an inpatient phase (phase 1) of 5 days, during which abstinence is achieved, followed by a 4 week outpatient phase (phase 2). A single infusion of ketamine or midazolam will occur on day 3 of Phase 1. In addition to measures of mindfulness and impulsivity, stress sensitivity tests are incorporated into the design in order to elucidate mechanisms of action. The study hypotheses are:

1. ketamine and MBRP will significantly increase the time to first use compared to placebo and MBRP in cocaine-dependent individuals.
2. ketamine and MBRP is significantly more likely to lead to abstinence from cocaine (no use over one week) as compared to placebo and MBRP.
3. ketamine and MBRP will significantly reduce subjective, endocrine, and physiological responses to stress (including cue exposure) as compared to placebo and MBRP.
4. ketamine and MBRP will significantly increase mindfulness, as assessed by the Five Facet Mindfulness Questionnaire (FFMQ), as compared to placebo and MBRP.

ELIGIBILITY:
Inclusion Criteria:

* Active cocaine dependence with at least 8 days of use or at least 4 binges of large amounts (>$200/occasion) over the past 30 days, and displaying at least one positive utox during screening
* Physically healthy
* No adverse reactions to study medications
* 21-60 years of age
* Capacity to consent and comply with study procedures, including sufficient proficiency in English
* Seeking treatment

Exclusion Criteria:

* Meets DSM IV criteria for current major depression, bipolar disorder, schizophrenia, any psychotic illness, including substance induced psychosis, and current substance-induced mood disorder with HAMD score > 12.
* Physiological dependence on another substance requiring medical management, such as alcohol, opioids, or benzodiazepines, excluding caffeine, nicotine, and cannabis
* Delirium, Dementia, Amnesia, Cognitive Disorders, or Dissociative disorders
* Current suicide risk or a history of suicide attempt within the past year
* Pregnant or interested in becoming pregnant during the study period
* Heart disease as indicated by history, abnormal ECG, previous cardiac surgery.
* Unstable physical disorders which might make participation hazardous such as end-stage AIDS, hypertension (>140/90), WBC < 3.5, active hepatitis or other liver disease with elevated transaminase levels (< 2-3 X upper limit of normal will be considered acceptable if PT/PTT is normal), renal failure (creatinine > 2, BUN >40), or untreated diabetes
* Previous history of ketamine or benzodiazepine misuse or abuse, and a history of an adverse reaction/experience with prior exposure to ketamine or benzodiazepine
* Recent history of significant violence (past 2 years)
* First degree relative with a psychotic disorder (bipolar disorder, schizophrenia, schizoaffective disorder, or psychosis NOS)
* BMI > 32, or a history of documented obstructive sleep apnea
* On psychotropic or other medications whose effect could be disrupted by participation in the study
* Patients who cannot comply with study procedures during the initial hospitalization phase

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Kleber, M.D., Study Chair — NYSPI; Elias Dakwar, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Dakwar E, Nunes EV, Hart CL, Foltin RW, Mathew SJ, Carpenter KM, Choi CJJ, Basaraba CN, Pavlicova M, Levin FR. A Single Ketamine Infusion Combined With Mindfulness-Based Behavioral Modification to Treat Cocaine Dependence: A Randomized Clinical Trial. Am J Psychiatry. 2019 Nov 1;176(11):923-930. doi: 10.1176/appi.ajp.2019.18101123. Epub 2019 Jun 24. PMID 31230464

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Midazolam
Started | 27 | 28
Completed | 27 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Midazolam | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (2) | 49 (1) | 47 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 22 | 19 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 20 | 34
  White | 5 | 2 | 7
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cocaine Use/Drop Out
Description: Number of participants who use cocaine and drop from study. During phase 2, patients will be assessed twice weekly by TLFB and urine toxicology for cocaine use. The day of first use will determine the length of time that transpired from discharge to the first lapse onto cocaine.
Time Frame: Over the four week period following discharge from the inpatient unit at Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 27 | 28
Participants | 16 | 26

2. Primary Outcome: Abstinence
Description: Abstinence is defined as 2 or greater weeks of no cocaine use, as ascertained by the TLFB and urine toxicology.
Time Frame: Abstinence will be assessed over 4 weeks starting at the last day of week 1 and continuing through the end of study at the last day of week 5
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 27 | 28
Participants | 13 | 3

ADVERSE EVENTS:
Time Frame: 5 weeks.
Arm/Group | Ketamine | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 3/27 | 7/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=27) | Midazolam (N=28)
sedation (Nervous system disorders) | 3 (3) | 7 (7) — sedation persisting for more than 1 hour post-infusion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes